CLINICAL TRIAL: NCT04616768
Title: A Feasibility Trial Using Remote Patient-reported Outcomes and Wearable Technology-reported Step Data to Compare Engagement, Utilization, and Functional Status in Patients With Incurable Lung and Gastrointestinal Cancers
Brief Title: PROStep: A Feasibility Trial Using PROs and Step Data to Monitor Patients With Lung and GI Cancers
Acronym: PROStep
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: UPCC 27921; 843616 (Other: UPenn IRB)
Record Dates: First submitted 2020-10-16; First posted 2020-11-05 (Actual); Results first posted 2025-07-02 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Cancer; Lung Cancer; Gastro-intestinal
Keywords: activity; patient-reported outcomes; GI
MeSH Terms: conditions — Neoplasms; Lung Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A - Control (No Intervention): An arm of ≤42 patients will not receive PRO surveys, a Fitbit device, or patient feedback texts messages. They will receive shortened utility surveys at 3 and 6 months following enrollment, but their clinicians will not receive dashboards or utility surveys.
- Arm B - Intervention without text feedback (Experimental): An arm of ≤42 patients enrolled intervention patients will be randomized to receive weekly patient-reported outcome questionnaires, be given Fitbits to monitor weekly step counts and utility surveys at 3 and 6 months following enrollment. Their clinicians will receive a "PROStep Dashboard" prior to their appointments and utility surveys at 3 and 6 months.
  Interventions: Other: PRO questionnaire; Other: Step monitoring; Other: PROStep Dashboard (clinicians)
- Arm C - Intervention with text feedback (Experimental): An arm of ≤42 patients enrolled intervention patients will be randomized to receive weekly patient-reported outcome questionnaires, be given Fitbits to monitor weekly step counts and utility surveys at 3 and 6 months following enrollment. Their clinicians will receive a "PROStep Dashboard" prior to their appointments and utility surveys at 3 and 6 months. Patients in this arm will receive an additional text prior to appointments that summarizes their symptoms and incorporates an active nudge question.
  Interventions: Other: PRO questionnaire; Other: Step monitoring; Other: Active nudge text feedback; Other: PROStep Dashboard (clinicians)

INTERVENTIONS:
Other: PRO questionnaire — These text message surveys will inquire about seven symptoms, requesting a response rating the patient's response. The seven symptoms have been selected by lung and GI oncology clinicians at PCAM from a list of twelve validated symptoms from the National Cancer Institute's Common Terminology Criteria for Adverse Events and will be scored on a five point scale from 0 (no present) to 4 (disabling). The patients will also receive a question asking about their activity level over the prior month
  Arms: Arm B - Intervention without text feedback; Arm C - Intervention with text feedback
Other: Step monitoring — A CRC will provide patients with a Fitbit at enrollment and instruct them on how to wear the Fitbit device and periodically sync the device with their phone which will send updated step data to the research team.
  Arms: Arm B - Intervention without text feedback; Arm C - Intervention with text feedback
Other: Active nudge text feedback — Intervention patients in arm c will receive text feedback describing worsening or severe symptoms collected from their remote PRO questionnaires (i.e. "Your following symptoms are severe or have gotten worse:") and their step count ("Your Fitbit step count compared to last week is worse."). They will also receive an "active nudge" question on their upcoming visit (i.e. "Do you plan on discussing these symptoms with your oncologist at your upcoming visit? Type "1" if you plan to discuss them; Type "2" if you do not plan to discuss them.").
  Arms: Arm C - Intervention with text feedback
Other: PROStep Dashboard (clinicians) — The study team will provide an updated PROStep Dashboard to lung or GI oncology clinicians for each patient enrolled in the intervention arms prior to their appointments. W2H will generate the dashboards and the study team will physically deliver it to their office or touchdown space or send electronically. The Dashboard will include:
  1. Home-based PRO report, including the weekly survey results for each question in tabular and graphical form
  2. Step data report, including a summary of number of daily steps in graphical form (with rolling weekly averages) and weekly averages in tabular form
  3. A list of all acute care utilization in the UPHS system in the prior 6 months including Oncology Evaluation Unit visits, Emergency department visits, Inpatient admissions
  4. Whether the patient has had an outpatient palliative care visit
  5. Whether the patient has had a documented Serious Illness Conversation
  Arms: Arm B - Intervention without text feedback; Arm C - Intervention with text feedback

SUMMARY:
Telemedicine allows clinicians to utilize modern telecommunication technology to provide healthcare services to patients including remote symptom monitoring. Given the spread of COVID-19 both locally and globally, is crucial to adapt accordingly in order to safely provide vulnerable cancer patient populations with optimal care while minimizing risk of exposure to COVID-19. In this study, the investigators will utilize remote monitoring of patients with cancer via weekly patient-reported outcome (PRO) collection through the Way to Health (W2H) smartphone application and step data through wearable Fitbit devices. Patients with incurable lung and gastrointestinal cancers will be recruited based on whether they receive their care in-clinic or remotely. They will respond to weekly phone-based symptom surveys and wear Fitbits that track step data. This data will be collated in a Palliative Care Assessment Dashboard (PROStep Dashboard) sent to clinicians prior to each oncology visit to help inform patient management. In this feasibility study, two arms of patients will be monitored with symptom surveys and Fitbits; the study will randomize these patients to either 1) receive text feedback or 2) receive no text feedback. A third arm of patients will be randomized to receive no feedback, symptom surveys, or Fitbit device. Clinicians for patients in each arm will receive the PROstep Dashboard. The study will determine feasibility of this monitoring approach, and compare patient adherence to symptom surveys and step data collection between the two intervention arms.

ELIGIBILITY:
Inclusion Criteria:

1. English-speaking
2. Have a diagnosis of incurable or Stage IV lung or gastrointestinal cancer
3. Receive primary oncology care with a thoracic or gastrointestinal medical oncology specialist at the Perelman Center for Advanced Medicine (i.e. does not have a local oncologist that provides cancer care, including other UPHS clinic sites)
4. Currently receiving or planned receipt within 2 weeks of IV chemotherapy (see exclusions below)
5. The patient has a smart phone that can receive SMS text messages and has blue-tooth capability that can connect to Fitbit.

Exclusion Criteria:

1. Age < 18 years
2. Patients has used a wheelchair, been bedbound or is unable to walk without assistance from other people every day for the past 7 days (patients are not excluded for the use of walkers or canes)
3. Patients who are receiving checkpoint inhibitor monotherapy or oral tyrosine kinase inhibitors
4. Patients who receive chemotherapy infusions at another UPHS site or outside of UPHS or whose primary oncologist is not in thoracic or gastrointestinal oncology groups at PCAM. Notably, patients who receive part of their chemotherapy regimen at home will still be allowed to enroll.
5. Lung cancer patients enrolled in an ongoing palliative care clinical trial that may lead to better communication regarding symptoms and functional status.
6. Clinician concerns about behavioral health issues that may prevent engagement with text message prompts
7. Are enrolled in another interventional clinical trial (as clinical trials often have a substantial symptom-reporting structure; non-interventional clinical trials are permitted e.g. trials that just involve blood tests)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Actual)
Dates: Start 2020-11-19 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ravi Parikh, MD, MPP, Principal Investigator — University of Pennsylvania
Locations (1):
- Perelman Center for Advanced Medicine (PCAM), Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Manz CR, Schriver E, Ferrell WJ, Williamson J, Wakim J, Khan N, Kopinsky M, Balachandran M, Chen J, Patel MS, Takvorian SU, Shulman LN, Bekelman JE, Barnett IJ, Parikh RB. Association of Remote Patient-Reported Outcomes and Step Counts With Hospitalization or Death Among Patients With Advanced Cancer Undergoing Chemotherapy: Secondary Analysis of the PROStep Randomized Trial. J Med Internet Res. 2024 May 17;26:e51059. doi: 10.2196/51059. PMID 38758583
- [Derived] Parikh RB, Schriver E, Ferrell WJ, Wakim J, Williamson J, Khan N, Kopinsky M, Balachandran M, Gabriel PE, Schuchter LM, Patel MS, Shulman LN, Manz CR. Remote Patient-Reported Outcomes and Activity Monitoring to Improve Patient-Clinician Communication Regarding Symptoms and Functional Status: A Randomized Controlled Trial. JCO Oncol Pract. 2023 Dec;19(12):1143-1151. doi: 10.1200/OP.23.00048. Epub 2023 Oct 10. PMID 37816198
- [Derived] Parikh RB, Ferrell W, Wakim J, Williamson J, Khan N, Kopinsky M, Balachandran M, Gabriel PE, Zhang Y, Schuchter LM, Shulman LN, Chen J, Patel MS, Manz CR. Patient and clinician nudges to improve symptom management in advanced cancer using patient-generated health data: study protocol for the PROStep randomised controlled trial. BMJ Open. 2022 May 12;12(5):e054675. doi: 10.1136/bmjopen-2021-054675. PMID 35551088

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm B - Intervention Without Text Feedback: An arm of ≤42 patients enrolled intervention patients will be randomized to receive weekly patient-reported outcome questionnaires, be given Fitbits to monitor weekly step counts and utility surveys at 3 and 6 months following enrollment. Their clinicians will receive a "PROStep Dashboard" prior to their appointments and utility surveys at 3 and 6 months.
  PRO questionnaire: These text message surveys will inquire about seven symptoms, requesting a response rating the patient's response. The seven symptoms have been selected by lung and GI oncology clinicians at PCAM from a list of twelve validated symptoms from the National Cancer Institute's Common Terminology Criteria for Adverse Events and will be scored on a five point scale from 0 (no present) to 4 (disabling). The patients will also receive a question asking about their activity level over the prior month
  Step monitoring: A CRC will provide patients with a Fitbit at enrollment and instruct them on how to wear the Fitbit device and periodically sync the device with their phone which will send updated step data to the research team.
  PROStep Dashboard (clinicians): The study team will provide an updated PROStep Dashboard to lung or GI oncology clinicians for each patient enrolled in the intervention arms prior to their appointments. W2H will generate the dashboards and the study team will physically deliver it to their office or touchdown space or send electronically.
- Arm C - Intervention With Text Feedback: An arm of ≤42 patients enrolled intervention patients will be randomized to receive weekly patient-reported outcome questionnaires, be given Fitbits to monitor weekly step counts and utility surveys at 3 and 6 months following enrollment. Their clinicians will receive a "PROStep Dashboard" prior to their appointments and utility surveys at 3 and 6 months. Patients in this arm will receive an additional text prior to appointments that summarizes their symptoms and incorporates an active nudge question.
  PRO questionnaire: These text message surveys will inquire about seven symptoms, requesting a response rating the patient's response. The seven symptoms have been selected by lung and GI oncology clinicians at PCAM from a list of twelve validated symptoms from the National Cancer Institute's Common Terminology Criteria for Adverse Events and will be scored on a five point scale from 0 (no present) to 4 (disabling). The patients will also receive a question asking about their activity level over the prior month
  Step monitoring: A CRC will provide patients with a Fitbit at enrollment and instruct them on how to wear the Fitbit device and periodically sync the device with their phone which will send updated step data to the research team.
  Active nudge text feedback: Arm C patients will receive a text describing worsening or severe symptoms collected from their remote PRO questionnaires and their step count and an "active nudge" question.
  PROStep Dashboard (clinicians)
Period: Overall Study
Arm/Group | Arm A - Control | Arm B - Intervention Without Text Feedback | Arm C - Intervention With Text Feedback
Started | 33 | 37 | 38
Completed | 31 | 24 | 25
Not Completed | 2 | 13 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A - Control | Arm B - Intervention Without Text Feedback | Arm C - Intervention With Text Feedback | Total
Number analyzed (Participants) | 33 | 37 | 38 | 108
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [51.8 to 65.2] | 59 [52 to 67] | 57 [51 to 65] | 59 [51.8 to 65.2]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 15 | 17 | 49
  Male | 16 | 22 | 21 | 59
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 1 | 3 | 1 | 5
  Race: Black or African American | 7 | 4 | 3 | 14
  Race: Other/Declined to identify | 0 | 0 | 2 | 2
  Race: White | 25 | 30 | 32 | 87
Symptoms [Count of Participants; unit: Participants]
  Poorly controlled | 3 | 2 | 5 | 10
  Well-controlled | 29 | 35 | 31 | 95
  Prefer not to answer | 1 | 0 | 2 | 3
Education [Count of Participants; unit: Participants]
  HS/GED | 6 | 7 | 7 | 20
  Some college | 4 | 2 | 4 | 10
  Vocational | 2 | 1 | 1 | 4
  Associate | 0 | 3 | 0 | 3
  Bachelor | 13 | 13 | 16 | 42
  Postgraduate | 8 | 11 | 10 | 29
Text Frequency [Count of Participants; unit: Participants] — Participants were asked "Generally, how often do you send/receive text messages?" on their enrollment questionnaire. Responses included: a. Not at all b. Fewer than 3 times weekly c. 3-5 times weekly d. Nearly every day e. Multiple times every day
  Participants
    3-5 times weekly | 0 | 3 | 0 | 3
    Nearly every day | 4 | 3 | 6 | 13
    Multiple times every day | 29 | 31 | 32 | 92

OUTCOME MEASURES:

1. Primary Outcome: Patient Perceptions of Symptom Management - How Well do You Feel Your Oncology Team Understands Your Symptoms (e.g. Nausea, Vomiting, Weight Loss, Etc.)?
Description: Patient utility surveys will use a 5-point Likert scale for responses scored 1-5. The two co-primary outcomes will compare the scores for the following two questions, measured at 6 months (or 3 months if the patient did not complete their 6 month survey), between intervention patients (Arms B + C) and control patients (Arm A).
  Likert scale responses are defined as: 1 = Not at all; 2 = Slightly; 3 = Moderately; 4 = Considerably; 5 = Completely.
Time Frame: These will be measured at 6 months after enrollment for each patient (or 3 months if the patient did not complete their 6 month survey)
Population: We originally were going to compare arms A v. B v. C, but due to lower-than-anticipated enrollment and higher-than-expected mortality, this was modified before the completion of the follow-up period and any data analysis to compare the control arm (A) with the combined intervention arms (B + C). The combined intervention was deemed to be more clinically relevant since we did not believe that responses to the symptom understanding question would be meaningfully different between Arms B and C.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Arm A: Control
- Arms B+C: Intervention
Arm/Group | Arm A | Arms B+C
Number analyzed (Participants) | 31 | 49
units on a scale | 4.5 (1) | 4.5 (1)

2. Primary Outcome: Patient Perception of Functional Status - How Well do You Feel Your Oncology Team Understands Your Activity Level and Ability to Function? (1-5)
Description: as for outcome 1
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A | Arms B+C
Number analyzed (Participants) | 31 | 49
units on a scale | 4.5 (.9) | 4.3 (1)

3. Secondary Outcome: Additional Analysis of the Primary Outcome Between Arms
Description: The following secondary outcome will compare the same questions measured at 3 months, between intervention patients (Arms B + C) and control patients (Arm A).
  * Q1 - How well do you feel your oncology team understands your symptoms (e.g. nausea, vomiting, weight loss, etc.)? (1-5)
  * Q2 - How well do you feel your oncology team understands your activity level and ability to function? (1-5)
  Likert scale responses are defined as: 1 = Not at all; 2 = Slightly; 3 = Moderately; 4 = Considerably; 5 = Completely.
Time Frame: These will be measured at 3 months after enrollment for each patient.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm A - Control | Arm B - Intervention Without Text Feedback | Arm C - Intervention With Text Feedback
Number analyzed (Participants) | 31 | 24 | 25
units on a scale
  Q1 | 4.5 (1) | 4.5 (1) | 4.4 (1.2)
  Q2 | 4.4 (.9) | 4.5 (.9) | 4.3 (1.1)

4. Secondary Outcome: Adherence
Description: We will compare cumulative adherence for patients in the intervention group (arm B and arm C). Each week, adherence will be defined as each week where the patient submits the weekly survey (i.e. adherence to PRO) and has step data for 4 of 7 days of the week (i.e. adherence to Fitbit platform), divided by the total number of weeks that the patient is enrolled in the trial.
  * Comparison of mean patient adherence at three months for patients in arm B vs arm C
  * Comparison of mean patient adherence at six months for patients in arm B vs arm C
Time Frame: Each patient will be enrolled in the trial for a total of six months.
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Number of Palliative Care Consults (Exploratory)
Time Frame: Each patient will be enrolled in the trial for a total of six months.
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Number of Documented Advanced Care Planning (ACP) Notes (Exploratory)
Time Frame: Each patient will be enrolled in the trial for a total of six months.
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Number of Documented Serious Illness Conversations (SIC) (Exploratory)
Time Frame: Each patient will be enrolled in the trial for a total of six months.
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Correlation Between Step, Heart Rate, Distance, Pace, Elevation and Sleep Data Trends, Patient Reported Outcomes, Patient and Clinician ECOG Assessment, and Patient Hospitalization and Survival (Exploratory)
Time Frame: Each patient will be enrolled in the trial for a total of six months.
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Patient Utility Surveys (Exploratory)
Description: The utility to patients is measured using survey data at 3 and 6 months. These use a 5-point Likert Scale (1-5). We will report descriptive statistics for this data (mean and standard deviation) followed by t-tests between each individual arm and between all intervention patients (Arms B + C) and control patients (Arm A).
Time Frame: Each patient will be surveyed at 3 and 6 months following enrollment.
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Clinician Utility Surveys (Exploratory)
Description: The utility to clinicians will be measured using survey data at three and six months. These similarly use a 5-point Likert scale (1-5) and we will report descriptive statistics for this survey data.
Time Frame: Each patient will be surveyed at 3 and 6 months following enrollment.
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Additional Analysis of the Primary Outcome Between Different Arms (6 Month) (Exploratory)
Description: The following exploratory outcomes will make the following comparisons for responses to the two questions in the primary outcomes:
  o Measured at 6 months (or 3 months if the patient did not complete their 6 month survey)
  * Between Arm B and Arm A
  * Between Arm C and Arm A
  * Between all Arms.
  Questions:
  * How well do you feel your oncology team understands your symptoms (e.g. nausea, vomiting, weight loss, etc.)? (1-5)
  * How well do you feel your oncology team understands your activity level and ability to function? (1-5)
  Likert scale responses are defined as: 1 = Not at all; 2 = Slightly; 3 = Moderately; 4 = Considerably; 5 = Completely.
Time Frame: These will be measured at 6 months (or 3 months if the patient did not complete their 6 month survey) after enrollment for each patient.
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Additional Analysis of the Primary Outcome Between Different Arms (3 Month) (Exploratory)
Description: The following exploratory outcomes will make the following comparisons for responses to the two questions in the primary outcomes:
  o Measured at 3 months
  * Between Arm B and Arm A
  * Between Arm C and Arm A
  * Between all Arms.
  Questions:
  * How well do you feel your oncology team understands your symptoms (e.g. nausea, vomiting, weight loss, etc.)? (1-5)
  * How well do you feel your oncology team understands your activity level and ability to function? (1-5)
  Likert scale responses are defined as: 1 = Not at all; 2 = Slightly; 3 = Moderately; 4 = Considerably; 5 = Completely.
Time Frame: These will be measured at 3 months after enrollment for each patient.
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 6 months
Description: CRC chart review
Arm/Group | Arm A - Control | Arm B - Intervention Without Text Feedback | Arm C - Intervention With Text Feedback
All-Cause Mortality (participants affected / at risk) | 1/33 | 7/37 | 2/38
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 0/33 | 0/37 | 0/38

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-10-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT04616768/Prot_SAP_000.pdf